CLINICAL TRIAL: NCT03547323
Title: A Randomized, Controlled, Open-label, Parallel Study in End Stage Renal Disease (ESRD) Patients on Hemodialysis to Determine Non-inferiority of the Theranova Dialyzer Compared to the FX80 Dialyzer
Brief Title: Study in End Stage Renal Disease (ESRD) Patients on Hemodialysis to Determine Non-inferiority of the Theranova Dialyzer Compared to the FX80 Dialyzer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0080002
Record Dates: First submitted 2018-05-16; First posted 2018-06-06 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theranova 400 Dialyzer (Experimental): One treatment session in an in-center setting.
  Interventions: Device: Theranova 400 Dialyzer
- FX80 Dialyzer (Active Comparator): One treatment session in an in-center setting.
  Interventions: Device: FX80 Dialyzer

INTERVENTIONS:
Device: Theranova 400 Dialyzer — An existing functioning vascular access (AVF, graft) must be in place and will be used for dialysis. Treatments will be administered by trained clinical staff. The use of temporary or tunneled dialysis catheters will not be allowed.
  Arms: Theranova 400 Dialyzer
Device: FX80 Dialyzer — An existing functioning vascular access (AVF, graft) must be in place and will be used for dialysis. Treatments will be administered by trained clinical staff. The use of temporary or tunneled dialysis catheters will not be allowed.
  Arms: FX80 Dialyzer

SUMMARY:
In China, the estimated prevalence of patients with ESRD receiving peritoneal dialysis (PD) or maintenance hemodialysis (HD) increased from 51.7 per million population (pmp) at the end of 2007 to 79.1 pmp at the end of 2008. There is a growing body of evidence that large uremic solutes play a significant role in clinical complications in dialysis patients. Since high-flux membranes show low permeability for large uremic solutes, extracorporeal blood purification treatments using these membranes have failed to significantly eliminate and reduce plasma levels of these molecules. To remove large sized uremic solutes by dialysis the membrane needs to have adequate permeability properties (pore size, porosity) for these solutes. The Theranova 400 contains a dialysis membrane that has a sharper sieving profile and a higher cutoff than that in conventional high-flux dialysis membranes. The primary objective of this study is to demonstrate non-inferiority of the Theranova Dialyzer compared to the FX80 with clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Patients able to give informed consent (IC) after an explanation of the proposed study.
* Patients who have Kt/Vurea > 1.2 for the last 2 measurements, where the most recent Kt/Vurea measurement is taken within 4 weeks before or during study screening.
* Patients with dialysis prescription (dialyzer, time, blood flow rate [QB], dialysis fluid flow rate [QD]) stable over 6 most recent treatments. The dialysis treatment duration time should be 3.5 - 4.5 hours per session, with QB of 220 - 300 mL/min and QD of 500 mL/min.
* Patients who are on stable anticoagulation prescription and dose.
* Patients with ESRD receiving chronic HD treatment with a history of thrice weekly HD, and at least 1 HDF session or HFHD, within 1 month prior to study.
* Patients must be stable on in-center HD and/or HDF for >3 months prior to study enrollment.
* Patients who have an adequate arteriovenous fistula (AVF) or graft, capable of providing a blood flow rate of at least 220 mL/min.

Exclusion Criteria:

* Patients who have acute renal failure with the chance for recovery.
* Patients who are pre-scheduled for a living kidney transplant within the next two months, who plan a change to PD within the next two months or who require single needle dialysis therapy.
* Pregnant and lactating women.
* Patients with positive serology tests for Hepatitis B surface antigen, positive Hepatitis C total antibody, HIV and syphilis.
* Patients with known hemodynamic instability, anemia (Hgb < 90 g/L), and/or severe bleeding risks secondary to coagulation disorders.
* Patients with active or ongoing infection per investigator's judgement.
* Patients with a history of solid tumors requiring anti-cancer therapy in the past or next 6 months or a life expectancy less than 1 year or patients with a history of a hematology neoplasm.
* Patients diagnosed with a NYHA Class IV congestive heart failure, or acute coronary syndrome and/or who have suffered a myocardial infarction within three months prior to the start of the study.
* Patients with a history of severe mental disorders.
* Patients who are currently participating or have previously participated in another interventional clinical trial in the past 4 weeks.
* Patients who have had an allergic response to polyarylethersulfone (PAES) or polsulfone membranes or have a history of poor tolerance to dialyzers with synthetic membranes.
* Patients with advanced liver, heart or pulmonary disease as judged by the Investigator.
* Patients with any comorbidity possibly conflicting with the study purpose or procedures as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Creatinine Clearance (K of Creatinine) | Up to 1 week
  One mid-week dialysis session
Urea Clearance (K of Urea) | Up to 1 week
  One mid-week dialysis session
Reduction Ratio (RR) of Beta-2 Microglobulin | Up to 1 week
  One mid-week dialysis session

SECONDARY OUTCOMES:
Kappa and Lambda Free Light Chains (FLCs) Reduction Ratio | Up to 1 week
  One mid-week dialysis session
Ultrafiltration Rate (QUF) | Up to 1 week
  One mid-week dialysis session
Urea reduction ratio (URR) | Up to 1 week
  One mid-week dialysis session

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Investigational Site, Beijing, Beijing Municipality
  - Investigational Site, Guangzhou, Guangdong
  - Investigational Site, Chengdu, Sichuan
  - Investigational Site, Hangzhou, Zhejiang